CLINICAL TRIAL: NCT05250089
Title: Performance of Emergency Physicians in the Management of Critical Situations Twenty-four Hours After the End of a Night Shift
Brief Title: Physicians Performance After Night Shifts
Acronym: URGENCE24
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/21/0241
Record Dates: First submitted 2022-01-11; First posted 2022-02-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Performance
Keywords: emergency; night shift; efficiency; physicians
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: single site prospective pilot study
Masking Description: The time frame of the simulation (post recovery or usual) will be unknown to the evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency physicians (Experimental): Each participant will have to carry out two simulation sessions. The first simulation will correspond to the "usual" evaluation, that is to say it will take place on a day that will not be preceded by night duty during the three previous nights.
  The second simulation will correspond to the assessment twenty-four hours after the end of a call, in the "post-recovery" period. The participant must therefore have performed a night shift the day before the day when the simulation takes place. This call must have a minimum duration of twelve hours on night shifts.
  Interventions: Other: Simulation

INTERVENTIONS:
Other: Simulation — Each simulation will focus on a trauma case deemed to be complex, that is to say one involving difficult decision-making. Each simulation session lasts approximately thirty minutes. It includes a time to complete the questionnaires necessary for carrying out the study, before and / or after the simulated practice depending on the type of questionnaire, a brief briefing on the simulation scenario, and the time for the simulated practice.

SUMMARY:
Emergency medicine is one of the professional activities integrating a night activity into working time. Concerns about the sleep deprivation that this activity generates have been growing for the past thirty years. However, at present, the pace - duration and repetition - of this activity does not yet seem to be optimized, and therefore continues to be the subject of questions in terms of safety of care and quality of life at work. One of the peculiarities of emergency medicine is that doctors have to work in a crisis situation. A situation is qualified as critical for a patient when his state of health is unstable, and with an evolution which can be rapidly pejorative. Crisis situations are at the heart of the emergency room profession, and due to their potential seriousness for the patients, it must be managed in all circumstances.

To cope with a crisis situation, a doctor needs to be efficient. However, performance calls for two types of skills: technical skills on one hand, and non-technical skills on the other.

This study therefore aims to answer the following question: are the non-technical skills of emergency physicians in the management of a crisis situation affected twenty-four hours after the end of a night shift? The study assesses the performance of emergency physicians via complex simulations at two time frames : 24h after a night shift (the post recovery performance simulation) and another time were the participant did not have night shifts in less than 3 nights (usual performance simulation).

DETAILED DESCRIPTION:
The study compare the post-recovery performance (PRP) and the usual performance (UP) of emergency physicians in the management of a critical situation. The PRP corresponds to the performance twenty-four hours after the end of a minimum 12 hours night shift, which corresponds to the usual time when a physician go back to work. The UP is defined as the performance achieved in the absence of night shifts during the three previous nights.

Each participants realises 2 complex simulations, each simulation will focus on a trauma case involving difficult decision-making. Each simulation session lasts approximately thirty minutes. It includes a time to complete the questionnaires necessary for carrying out the study, before and / or after the simulated practice depending on the type of questionnaire, a brief interview on the simulation scenario, and the time for the simulated practice.The simulation environment of the study is as close as possible to a reception room for vital emergencies (SAUV), in order to be as close as possible to the usual professional environment of the participants.

During the simulated practice, a technician manages the progress of the scenario under the supervision of an emergency doctor controlling it. In the room, each participant is accompanied by two trained paramedics, whose roles will depend on the scenarios.

The performance is assessed via the Ottawa Crisis Resource Management Global Rating Scale (Ottawa GRS), questionnaires and an electrocardiogram (ECG).

ELIGIBILITY:
Inclusion Criteria:

* be an emergency doctor with an emergency medicine capacity,
* work full time in the emergency medicine center of the Toulouse University Hospital
* on call in at least one of the emergency reception services of the Toulouse University Hospital
* to have given his non-opposition to participate and his authorization of right to his image and his voice within the framework of the research

Exclusion Criteria:

* non-emergency doctor
* emergency doctor not on call in at least one of the emergency services of the Toulouse University Hospital
* professional with a declared personal or professional conflict with one of the members of the group

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
non-technical efficiency via the Ottawa GRS | 24 hours after a night shift
  Overall non-technical skill score assessed using the Ottawa Crisis Resource Management Global Rating Scale (Ottawa GRS).
  The Ottawa GRS scale assesses the following five criteria:
  * leadership skills
  * situational awareness
  * communication skills
  * problem solving
  * resource management For each of the criteria, a score between 1 and 7 is attributed. The scoring is made as follows: a score of 1 corresponds to a novice performance, a score of 3 corresponds to a performance of a novice with experience in Crisis Resource Management (CRM) and resuscitation, a score of 5 corresponds to the performance of a physician with sufficient experience in CRM and resuscitation to properly manage a crisis situation, finally a score of 7 corresponds to the performance of a physician expert in CRM and resuscitation.
  An average score of the five scores is taken to obtain an overall proficiency score, also out of 7, which will be used to compare Post Recovery Performance and Usual Performance
non-technical efficiency via the Ottawa GRS | after a minimum of 3 nights free of night work
  Overall non-technical skill score assessed using the Ottawa Crisis Resource Management Global Rating Scale (Ottawa GRS).
  The Ottawa GRS scale assesses the following five criteria:
  * leadership skills
  * situational awareness
  * communication skills
  * problem solving
  * resource management For each of the criteria, a score between 1 and 7 is attributed. The scoring is made as follows: a score of 1 corresponds to a performance judged to be that of a novice, a score of 3 corresponds to a performance of a novice with experience in CRM and resuscitation, a score of 5 corresponds to the performance of a physician with sufficient experience in CRM and resuscitation to properly manage a crisis situation, finally a score of 7 corresponds to the performance of a physician expert in CRM and resuscitation.
  An average score of the five scores is taken to obtain an overall proficiency score, also out of 7, which will be used to compare Post Recovery Performance and Usual Performance

SECONDARY OUTCOMES:
Physiologic stress | 24 hours after a night shift
  Comparison of the psychological stress of emergency physicians during a simulated critical situation, between post-recovery time frame and usual time frame.
  Physiological stress will be assessed via the measurement of heart rate variability, thanks to the analysis of data from a Holter ECG worn by the participant during each simulated practice (Post Recovery Performance and Usual Performance).
Physiologic stress | after a minimum of 3 nights free of night work
  Comparison of the psychological stress of emergency physicians during a simulated critical situation, between post-recovery time frame and usual time frame.
  Physiological stress will be assessed via the measurement of heart rate variability, thanks to the analysis of data from a Holter ECG worn by the participant during each simulated practice (Post Recovery Performance and Usual Performance).

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Henri HOUZE-CERFON, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No